CLINICAL TRIAL: NCT01801241
Title: Comparison of Glenoid Component Position Using Intelligent Reusable Instrument (IRI) vs Standard Surgical Instruments
Acronym: IRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Joseph Iannotti, Cheif of Staff, Executive Administration Florida, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPP-12-245
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Anatomic Total Shoulder Arthroplasty
Keywords: Anatomic total shoulder arthroplasty; Glenoid; Patient specific information; Computer simulation; Computer assisted tomography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Anatomic TSA using SOC Instrumentation (Active Comparator): During Anatomic Total Shoulder Arthroplasty, the surgeon will use the pre operative CT scan at least two weeks prior to surgery to define the glenoid pathology, select the implant of choice and plan the placement of that implant in the desired position. This information will be available to the surgeon at the time of surgery but the SmartBone models and the IRI will not be available. The surgeon will have pre operative x-rays and the pre operative CT scan provided by the radiology department for intra - use. The surgeon will perform the surgery using any of the instruments provided for guide pin placement operative the. These include a wide variety of free hand and adjustable guides that assist the surgeon for placement of the guide pin for location and trajectory.
  Interventions: Procedure: Anatomic Total Shoulder Arthroplasty
- Anatomic TSA Using IRI Instrumentation (Experimental): During Anatomic Total Shoulder Arthroplasty, the surgeon will have use of the SmartBone model of the patient's anatomy and glenoid guide-pin location, and the Intelligent Reuseable Instrument for placement of the glenoid implant.
  Interventions: Device: Anatomic TSA using IRI Instrumentation; Procedure: Anatomic Total Shoulder Arthroplasty

INTERVENTIONS:
Device: Anatomic TSA using IRI Instrumentation — Anatomic Total Shoulder Arthroplasty (TSA) will be performed using the SmartBone and Intelligent Reusable Instrument (IRI) to transfer the pre-operative plan for glenoid implant positioning to the patient's anatomy.
  Arms: Anatomic TSA Using IRI Instrumentation
Procedure: Anatomic Total Shoulder Arthroplasty — Anatomic Total Shoulder Arthroplasty will be performed by the two surgeons of the study as their Standard of Care. All procedures associated with the surgery will be the same in the two arms, with the exception of the tools used to place the guide pin for placement of the glenoid implant.

SUMMARY:
The proposed clinical study will enroll patients indicated for standard of care anatomic total shoulder arthroplasty. They will receive all pre operative testing, intra-operative care including all implants and post operative care that is standard of care and specific to the surgeon and patients decisions for care. The only difference between the study groups will be the type of surgical instruments used to place the glenoid guide pin. In all cases the surgeon is able and allowed to use their own surgical judgment to place the guide pin, prepare the bone and place the desired implant. In cases that are randomized to the IRIS group the surgeon can use any and all of the standard instruments or guides provided by the implant manufacturer as the surgeon would use in the group of patients randomized to the standard surgical group. If the surgeon chooses not to use the IRIS instruments then this would be noted as a deviation in plan, the reasons recorded and the patient would be excluded from the study without post operative imaging and there pre - operative and intra - operative data would be analyzed for the purpose of understanding the reasons for failure of the IRIS technology to provide surgical assistance for guide pin placement. For patients included in the post operative data analysis will a study specific shoulder CT scan prior to discharge from the hospital to assess the position of the implant. Deviation in the location and position of the implant as compared plan will be our primary outcome measure. Investigators will compare difference between technologies, differences within and between surgeons and the influence of the severity of the pre operative pathology on the two methods of surgical care.

DETAILED DESCRIPTION:
The study will enroll 60 patients into a randomized clinical trial, 30 in the standard of care surgery group and 30 in the IRI surgical group. Investigators will have two surgeons with experience in shoulder arthroplasty and the IRIS and SmartBones technology. Investigators will require a minimum of ten patients in each surgical group (n=20) from any one surgeon. Enrollment by any one surgeon will be limited so that all surgeons achieve a minimum of 20 cases enrolled. All patients will have the standard of care indications for an anatomic total shoulder arthroplasty and will give informed consent for both the surgery and participation in this study. Consent and enrollment will be obtained by the surgeon during a routine office evaluation. All patients will get standard of care pre operative x-rays and CT scan at least three weeks prior to surgery. Scan quality must meet study specific criteria and we expect but will not require that the scans will be performed at the Cleveland Clinic. The pre operative CT scan will be placed within the investigators' pre operative planning software (OrthoVis Cleveland Clinic). The surgeon will use this software to assess the glenoid bone pathology and select the optimal implant and placement of that implant. After pre operative planning each patient will be randomized into either an IRIS group which will use the pre-operative 3D surgical planning software and the data from this software to create a sterile SmartBone model containing the desired location of the glenoid guide pin and instructions for use of an intelligent reusable instrument to assist the surgeon in placement of the guide pin within the patient's glenoid. In the standard treatment group the surgeon will receive the data from the pre operative surgical simulation and use the instruments provided by the implant manufacturer. Statistician provided randomization envelopes will be provided to sort the patients into experiment and standard of care groups.

Patients will have standard of care indications for primary anatomic arthroplasty and be able to get a pre-operative shoulder CT scan at the Cleveland Clinic or at an outside facility so long as the study includes the entire scapula and has 1mm or thinner sections. These parameters are required for accurate pre operative planning as well as comparison with the post operative CT scans. Standard of care pre- and post-operative x-rays (AP and axillary views) will also be obtained and can be preformed at the Cleveland Clinic or acquired from another health care facility. In all patients the standard x-rays and CT images provided by the radiology department will be available to the surgeon before and during the surgery.

For the experimental group, the cannulated IRIS instrument designed for glenoid pin placement is placed over the guide wire that is contained within the sterile SmartBone and the legs of the instrument are adjusted to record the relationship (location and trajectory) of the guide pin in relation to the patient specific glenoid anatomy. This is done at the time of surgery to properly mimic the desired pin placement. The location of each leg of the IRI is marked on the SmartBone with a surgical pen. The instrument is then removed from the smart bone model. The SmartBone model is visually compared by the surgeon to the exposed bone surface to ensure that the two match for shape and size. Any adjustments to the surgical site may be done by the surgeon to optimize the match between the model and the exposed glenoid surface. The marks placed by the surgeon on the model are then transferred to the patient bone using a surgical marker or bovie. These marks are in a general location as determined by the surgeon and assist in the placement of the IRI. The IRI is placed onto the patient bone surface in the same manner as it was placed on the SmartBone model and a guide pin provided by the manufacturer is placed into the desired position. The surgeon then removes the IRI and compares by visual inspection the location and trajectory of the guide pin in relation to the patients bone surface and that within the SmartBone's model. Any adjustments in guide pin position can be performed by the surgeon based upon surgical judgment. The surgeon can make any change needed and use any means or instrument that would otherwise be used for standard of care surgery to place the guide pin in any position that the surgeon believed to be best for the patient. If the pin is changed without the use of the IRI then the patient will be excluded from this study and the reasons for failure of the IRI technology to provide accurate pin placement based upon the surgeon's sole determination of accuracy will be recorded and later analyzed as a failure to treat. These patients will not receive post operative CT Scans as we would not be able to use the data within any one group as defined by this study. After placement of the guide pin the remainder of the procedure is completed in the same manner for both groups, using the implant manufacturer's equipment.

In the standard instrument group the surgeon will use the pre operative CT Scan at least two weeks prior to surgery to define the glenoid pathology, select the implant of choice and place that implant in the desired position. This information will be available to the surgeon at the time of surgery but the SmartBone models and the IRI will not be available. The surgeon will have the pre operative x-rays and the pre operative CT scan provided by the radiology department for intra - operative use. The surgeon will perform the surgery using any of the instruments provided for guide pin placement. These include a wide variety of free hand and adjustable guides that assist the surgeon for placement of the guide pin for location and trajectory. Which tools are used for each case will be recorded at the time of surgery.

Prior to discharge, the patient will receive a post-operative CT scan. This will be a CT scan performed with the patient's arm by the side in a supine position using metal artifact reduction techniques. In addition patients will receive a second CT scan performed 1 year (± 1 month) from surgery. These scans will be performed with the patient in the lateral decubitus position with their arm in the overhead position again using metal artifact reduction techniques. The second set of images produced with a different body and arm position will generate much less metal artifact than those obtained immediately after surgery. This position can not be safely obtained until 3- 6 months after surgery and requires healing of the tissues and rehabilitation of the shoulder. We have shown that in a small number of patients the glenoid component can shift in position within the first 3-6 months after surgery making the first CT scan more accurate for implant position. The images obtained from the post-operative CT scans are placed back into the surgical software and the 3D reconstruction of the post-operative scapula with the implants is compared to the pre-operative plan. Using measurement tools within the software, developed at the Cleveland Clinic, we will compare the position of the actual glenoid component placed in the patient with the desired position specified by the plan. The use and validation of these imaging methods to precisely measure implant position has been performed at the Cleveland Clinic in a prior IRB approved clinical trial (IRB 10-582).

The participating surgeons will be Dr. Joseph Iannotti and Dr. Eric Ricchetti.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion, a primary anatomic total shoulder arthroplasty must be indicated for the patient.

Exclusion Criteria:

* Age less than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Iannotti, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Orthopaedic and Rheumatologic Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IDP with other researchers.

REFERENCES:
- [Background] Hendel MD, Bryan JA, Barsoum WK, Rodriguez EJ, Brems JJ, Evans PJ, Iannotti JP. Comparison of patient-specific instruments with standard surgical instruments in determining glenoid component position: a randomized prospective clinical trial. J Bone Joint Surg Am. 2012 Dec 5;94(23):2167-75. doi: 10.2106/JBJS.K.01209. PMID 23224387
- [Derived] Iannotti JP, Weiner S, Rodriguez E, Subhas N, Patterson TE, Jun BJ, Ricchetti ET. Three-dimensional imaging and templating improve glenoid implant positioning. J Bone Joint Surg Am. 2015 Apr 15;97(8):651-8. doi: 10.2106/JBJS.N.00493. PMID 25878309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anatomic TSA Using SOC Instrumentation | Anatomic TSA Using IRI Instrumentation
Started | 29 | 27
Completed | 21 | 25
Not Completed | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anatomic TSA Using SOC Instrumentation | Anatomic TSA Using IRI Instrumentation | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 8 | 12 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Difference in Glenoid Component Placement (Inclination and Version)
Description: The overall difference in component placement between standard of care instrumentation and intelligent reusable instrumentation will be compared (Inclination and Version).
  Inclination: the angle measurement of the position of the glenoid surface or glenoid implant in the superior-inferior direction. Version: the angle measurement of the position of the glenoid surface or glenoid implant in the anterior-posterior direction.
Time Frame: Two weeks post surgery
Measure: Mean (95% Confidence Interval); unit: degree
Arm/Group | Anatomic TSA Using SOC Instrumentation | Anatomic TSA Using IRI Instrumentation
Number analyzed (Participants) | 21 | 25
degree
  Inclination | 4.1 [2.7 to 5.5] | 3.1 [2.1 to 4.2]
  Version | 4.3 [3.1 to 5.5] | 4.0 [3.0 to 5.1]

2. Primary Outcome: Difference in Glenoid Component Placement (AP and SP).
Description: The overall difference in component placement between standard of care instrumentation and intelligent reusable instrumentation will be compared (Anteroposterior position and Superoinferior position).
Time Frame: Two weeks post surgery
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Anatomic TSA Using SOC Instrumentation | Anatomic TSA Using IRI Instrumentation
Number analyzed (Participants) | 21 | 25
mm
  Anteroposterior position | 1.7 [1.2 to 2.2] | 1.1 [0.8 to 1.5]
  Superoinferior position | 1.5 [0.9 to 2.2] | 0.9 [0.5 to 1.3]

3. Secondary Outcome: Difference in Glenoid Component Position Within and Between Surgeons
Description: Investigators will compare the placement of the glenoid component between the two technologies within and between the two surgeons.
Time Frame: Two weeks post surgery
Population: Outcome measures data not collected/ no patients analyzed for this OM. A broader study including different surgeons is required to test the effectiveness of this technology.
Arm/Group | Anatomic TSA Using SOC Instrumentation | Anatomic TSA Using IRI Instrumentation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Effect of Severity of Shoulder Pathology
Description: Investigators will evaluate the difference in glenoid component position between SOC and IRI technologies based on severity of shoulder pathology (using Walch classifications), if the difference between the severity of shoulder pathology is less than p-value 0.05. If p-value is greater than 0.05, investigators will not evaluate the difference in the glenoid component position between SOC and IRI.
Time Frame: Two weeks post surgery
Population: The Walch classification of glenoid morphology is the most commonly used system describing glenohumeral pathology in primary osteoarthritis. Glenoids were classified as asymmetric moderate-to severe posterior glenoid bone loss (Walch type-C or moderate to-severe type-B2 and B3 glenoids), without bone loss (Walch type-A1 glenoid), posterior bone loss requiring <10 degrees of correction (Walch type-B1 or mild type-B2 and B3 glenoids), or symmetric glenoid bone loss (Walch type-A2 glenoid).
Measure: Count of Participants; unit: Participants
Arm/Group | Anatomic TSA Using SOC Instrumentation | Anatomic TSA Using IRI Instrumentation
Number analyzed (Participants) | 21 | 25
Participants
  A1 | 4 | 3
  A2 | 7 | 5
  B1 | 2 | 2
  B2 | 6 | 12
  C | 2 | 3
Statistical Analysis 1: Comparison: Anatomic TSA Using SOC Instrumentation vs Anatomic TSA Using IRI Instrumentation; Test type: Superiority; p = 0.45, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Approximately one year from the time of surgery.
Description: Adverse events include excessive bleeding, infection, fracture nerve injury or need for revision surgery during the term of this study which is expected to be approximately one year from the time of surgery. All-cause mortality was not monitored/assessed for this study.
Arm/Group | Anatomic TSA Using SOC Instrumentation | Anatomic TSA Using IRI Instrumentation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/25
Other Adverse Events (participants affected / at risk) | 0/21 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT01801241/Prot_SAP_000.pdf